CLINICAL TRIAL: NCT02799693
Title: Outcomes of Intramural Needle Ablation for Recurrent Ventricular Tachycardia That Has Failed Conventional Radiofrequency Ablation
Brief Title: Intramural Needle Ablation for Ventricular Tachycardia
Status: Completed | Type: Observational
Sponsor: John Sapp (Other)
Responsible Party: Sponsor-Investigator, John Sapp, MD FRCPC FRHS, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: Sapp002
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Ventricular Tachycardia
Keywords: Catheter Ablation; Ventricular Tachycardia; Intramural Needle Catheter
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recurrent VT failing RF ablation: Patients undergoing intramural needle catheter ablation of recurrent monomorphic ventricular tachycardia who have failed prior attempted radiofrequency catheter ablation.

SUMMARY:
This is a single-arm non-randomized prospective observational cohort study to assess the outcomes of patients undergoing intramural needle catheter ablation of recurrent ventricular tachycardia that has failed antiarrhythmic drug therapy and standard radiofrequency (RF) catheter ablation. Following ablation, patients will be monitored for 6 months. The duration of the study is up to 4 years.

DETAILED DESCRIPTION:
This is an observational prospective cohort study of patients undergoing needle catheter ablation. Patients with recurrent sustained or incessant ventricular tachycardia who have recurrent monomorphic ventricular tachycardia that has failed antiarrhythmic drug therapy and prior catheter ablation who are undergoing intramural needle ablation for VT will be offered participation. Data will be collected during the procedure and during follow-up. Patients will be monitored in hospital for complications and during 6 months follow-up.

Data Collection:

Baseline Data: Baseline demographic information and a narrative medical history will be collected on all patients, including documentation of prior cardiac history, and arrhythmia history, as well as prior medications and cardiac procedures.

Procedural data: Details of the procedure including both procedural methods and arrhythmias induced, ablation parameters, needle deployments, recordings and response to procedure.

Followup data: Adverse events will be collected for events which are documented during enrollment and follow-up. During follow-up, hospitalizations will be collected, need for further procedures, implantable defibrillator therapies and procedures will be collected, as well as follow-up echocardiography findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing catheter ablation using the needle ablation catheter for ventricular arrhythmias.

Exclusion Criteria:

* Patient refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with recurrent ventricular tachycardia who have failed radiofrequency catheter ablation who are undergoing intramural needle catheter ablation procedures.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Freedom from hospitalization for recurrent VT during 6 months following ablation | 6 months
  Control of VT as defined by: freedom from hospitalization for recurrent VT during the 6 months following ablation
Absence of serious adverse events attributable to the procedure which occur within 30 days of the ablation procedure | 6 months
  Absence of all serious adverse events that are potentially procedure related and occur within 30 days of the ablation procedure.

SECONDARY OUTCOMES:
Acute Procedural Success | 6 hours
  Termination of at least one clinical or presumptive clinical monomorphic VT by RF ablation or rendering that VT no longer inducible
Acute procedural complications | 24 hours
  Any complications occurring within 24 hours post procedure described as probably or possibly related to the VT catheter ablation procedure
Number of inducible VT morphologies | 6 hours
  Number of VT morphologies induced during catheter ablation
ICD therapy - shocks | 3 months
  Number of VT events treated with appropriate ICD shocks at 3 months post procedure
ICD therapy - shocks | 6 months
  Number of VT events treated with appropriate ICD shocks at 6 months post procedure
ICD therapy - ATP | 3 months
  Number of VT events treated with antitachycardia pacing (without shock) during 3 months follow-up post-ablation procedure
ICD therapy - ATP | 6 months
  Number of VT events treated with antitachycardia pacing (without shock) during 6 months follow-up post-ablation procedure
ICD Therapy | 3 months
  Number of VT events treated with antitachycardia pacing (with shock) during 3 months follow-up post-ablation procedure
ICD Therapy | 6 months
  Number of VT events treated with antitachycardia pacing (with shock) during 6 months follow-up post-ablation procedure
VT storm | 3 months
  Number of VT storm events during 3 months follow-up
VT storm | 6 months
  Number of VT storm events during 6 months follow-up
VT events | 3 months
  Difference in number of VT events during 3 months prior to and following procedure
VT events | 6 months
  Difference in number of VT events during 6 months prior to and following procedure
Recurrent VT | 6 months
  Time to first recurrent VT
Appropriate ATP | 6 months
  Time to first appropriate ATP
Appropriate ICD shock | 6 months
  Time to first appropriate ICD shock
VT Storm | 6 months
  Time to first VT storm
Antiarrhythmic Drug Therapy | 6 months
  Changes in antiarrhythmic drug therapy post-procedure
Total appropriate ICD shocks | 3 months
  Total number of appropriate ICD shocks during 3 months follow up
Total appropriate ICD shocks | 6 months
  Total number of appropriate ICD shocks during 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: John Sapp, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No